CLINICAL TRIAL: NCT04187651
Title: Use of Platelet Rich Plasma in Treatment of Perianal Fistula
Brief Title: PRP Use in Treatment of Fistula Ano
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Barış Sevinç, Assoc. Prof., Uşak University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRPF
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Fistula in Ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: PRP gel will be applicated to all cases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP gel application (Experimental): PRP application for perianal fistula
  Interventions: Other: platelet rich plasma

INTERVENTIONS:
Other: platelet rich plasma — platelet rich plasma prepared from the patients' own blood will be applied to the fistula tract

SUMMARY:
In treatment of perianal fistula several methods are described. However, since the Hippocrates basics of surgical treatment has not changed very much. the aim of this study is to evaluate the effectiveness of PRP gel in treatment of perianal fistula.

DETAILED DESCRIPTION:
Perianal fistula is a chronic condition that seriously affects the patients' quality of life. There are different treatment modalities used in treatment. Recently sphincter preserving methods are becoming more popular with low complication rates. Most of this methods aiming the closure of fistula tract by different pathways.

Platelet rich plasma (PRP) is used in a wide range of conditions in medicine. The investigator's team showed the effective treatment of pilonidal disease by use of PRP gel. In the recent study, aim to evaluate the effectiveness of PRP gel in treatment of perianal fistula.

Patients with perianal fistula will be evaluated for the study. After taking permission with informed consent; cases will be included in the study. Cases with inflammatory bowel disease, platelet function disorders or connective tissue disorders that may alter wound healing will be excluded from the study.

After, PRP application to the fistula tract patients will be taken to follow up. Perianal fistulas will be followed by magnetic resonance imaging 1 month after the application. Pre-application and post-application scans will be used for the evaluation of the treatment success.

ELIGIBILITY:
Inclusion Criteria:

* patients with perianal fistula
* signing the informed consent form
* above the age of 18

Exclusion Criteria:

* inflammatory bowel disease
* previous radiation therapy
* having connective tissue disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
percentage of the cure rate | 1 month
  closure of the fistula tract will be evaluated by physical examination and magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Barış Sevinç, M.D., Principal Investigator — Uşak University Medical School
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No